CLINICAL TRIAL: NCT03804294
Title: Effect of Vitamin D on Outcome of Assisted Reproductive Technology(ART)
Brief Title: Effect of Vitamin D on Outcome of Assisted Reproductive Technology(ART);
Acronym: ART
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Peking University Third Hospital (Other)
Responsible Party: Principal Investigator, Zhi Xu, associate professor, Peking University Third Hospital
Other Study IDs: Vitamin D and ART
Record Dates: First submitted 2019-01-11; First posted 2019-01-15 (Actual); Last update posted 2019-01-17 (Actual); Status verified 2019-01

CONDITIONS: ART

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — serum
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- vitamin D-ART: Infertile couples who undergo their ﬁrst IVF/ICSI and IUI cycle in Reproductive Medicin Center of Peking university Third Hosiptal.

SUMMARY:
Vitamin D has many biological functions. Vitamin D receptors are widely distributed in the male and female reproductive system. Animal experiments have shown that vitamin D deficiency can affect hormone synthesis and gamete formation, reduce sperm motility, and may be related to diseases such as PCOS and endometriosis. Population studies suggest that vitamin D may be related to androgen levels and sperm quality, but whether vitamin D affects the outcome of assisted reproduction is controversial and inconclusive. This study intends to explore whether vitamin D affects the outcome of assisted reproduction through a large sample cohort study.

DETAILED DESCRIPTION:
Vitamin D plays an important role in reproduction, while there is high prevalence of vitamin D deficiency. Serum 25(OH)D was categorized according to clinically accepted ranges for vitamin D deﬁciency (<20 ng/mL), insufﬁciency (20-30 ng/mL), and replete (>30 ng/mL).

This is a retrospective cohort study of about 2000 infertile couples who undergo their ﬁrst IVF/ICSI and IUI cycle at Reproductive Medicine Center of Peking University Third Hospital. Patients will be excluded if they refuse to be recruited. Serum samples are collected the day when patients first time to Reproductive Medicine Center and were stored at -20℃ until assayed. Life style of patients is collected by questionair. Vitamin D status is measured by assessing circulating levels of 25(OH)D in frozen, never previously thawed serum samples using radioimmunoassay.

The investigators will comapere the ART outcomes in different groups according to serum 25(OH)D status.

In female, the primary outcome is clinical pregnancy rates deﬁned as the presence of an intrauterinesac with an embryonic pole demonstrating cardiacactivity at 7 weeks of gestation. Secondary outcomes are quality of embryo, positive hCG rates and live birth rates.

In male, the primary outcome is semen quality, such as semen volume, sperm concentration, sperm motility, morphologically normal percent and progressive motile spermatozoa percent. Secondary outcomes are clinical pregnancy rates and live birth rates.

ELIGIBILITY:
Inclusion Criteria:

infertile couples who undergo their ﬁrst IVF/ICSI and IUI cycle at Reproductive Medicine Center of Peking University Third Hospital.

Exclusion Criteria:

refusing to be recruited.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: infertile couples
Sampling Method: Probability Sample
Enrollment: 4000 (Estimated)
Dates: Start 2018-11-28 (Actual); Primary Completion 2019-12-01 (Estimated); Study Completion 2020-07-01 (Estimated)

PRIMARY OUTCOMES:
clinical pregnancy rates | 12 weeks after transplantation
  Time Frame:
  the presence of an intrauterinesac with an embryonic pole demonstrating cardiacactivity

CONTACTS AND LOCATIONS:
Overall Officials: XU ZHI, Study Chair — Peking University Third Hospital
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Chen Y, Liu D, Zeng L, Xu H, Jiang H, Yang R, Wang H, Yan L, Li R, Qiao J, Zhi X. Effect of serum 25-hydroxyvitamin D levels on sperm quality and assisted reproductive technology outcomes for men of infertile Chinese couples. Andrology. 2020 Sep;8(5):1277-1286. doi: 10.1111/andr.12818. Epub 2020 Jun 3. PMID 32412142